CLINICAL TRIAL: NCT00198484
Title: Evaluation of Vitrase (Hyaluronidase for Injection) Ovine, 200 USP Units/mL, as an Adjuvant to Increase the Absorption and Dispersion of Other Injected Drugs Prior to Ocular Surgery
Brief Title: Evaluation of Vitrase as a Spreading Agent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISTA-VIT-SA-CS06
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Pain
Keywords: Adjuvants, Anesthesia; Spreading Factor
MeSH Terms: conditions — Pain | interventions — Chondroitinases and Chondroitin Lyases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitrase (Experimental): ovine hyaluronidase injection 150 USP Units in 1 mL solution. Single dose of Vitrase will be administered as an adjuvant prior to ophthalmologic surgery
  Interventions: Drug: Vitrase

INTERVENTIONS:
Drug: Vitrase
  Other Names: ovine hyaluronidase

SUMMARY:
The purpose of this study is to determine whether Vitrase (hyaluronidase for injection) is effective as a spreading agent for other injected drugs prior to ocular surgery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an ophthalmic surgical procedure

Exclusion Criteria:

* Documented history of hypersensitivity to hyaluronidase or any other ingredient in Vitrase
* Known history of hypersensitivity reaction to bee or wasp venom
* Needing enhanced absorption and dispersion of dopamine, alpha agonist drugs, furosemide, the benzodiazepines, or phenytoin
* Inflammation or apparent clinical signs of infection in the area where Vitrase was to be injected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-10; Primary Completion 2004-12 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Physician Satisfaction Survey | 1-2 days
  Physician evaluation of effectiveness of Vitrase as an adjuvant and overall satisfaction, via questionnaire;

SECONDARY OUTCOMES:
Adverse Events | 1-2 days
  occurrence, severity, relationship, duration, resolution, and seriousness of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Grillone, PhD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (18):
- United States (18):
  - David Wirta, MD, Inc., Newport Beach, California
  - Richard A Lewis, MD, Sacramento, California
  - E Randy Craven, MD, Littleton, Colorado
  - The Eye Care Group, New Haven, Connecticut
  - Advanced Eye Care, PC, Fort Oglethorpe, Georgia
  - Donald E Beahm, MD, Great Bend, Kansas
  - Cincinnati Eye Institute NKY, Edgewood, Kentucky
  - Cornea Consultants, Boston, Massachusetts
  - Hunkeler Eye Institute, Kansas City, Missouri
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - David L Schwartz, MD, Tulsa, Oklahoma
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Texan Eye Care PA, Austin, Texas
  - Ophthalmology Service, Brooke Army Medical Center, Fort Sam Houston, Texas
  - Ophthalmology Visual Science, Galveston, Texas
  - Houston Eye Associates, Houston, Texas
  - David G Shulman, MD, San Antonio, Texas
  - Central Texas Eye Center, San Marcos, Texas